CLINICAL TRIAL: NCT07280715
Title: Digital Remote Patient Monitoring and Triage During Cancer Immunotherapy
Brief Title: Investigating Real-Time Immunotherapy Symptoms Study
Acronym: IRIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Carissa Low, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY25090094
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Melanoma (Skin Cancer); Immunotherapy
Keywords: quality of life; adverse events
MeSH Terms: conditions — Neoplasms; Melanoma

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the digital remote monitoring group or usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital remote monitoring group (intervention) (Experimental): Participants will complete baseline, midpoint, and end of study measures and complete the Short Physical Performance Battery (SPPB) as feasible. Participants will rate symptoms weekly for 90 days using PRO-CTCAE questions to assess symptoms commonly associated with immune-related adverse events (irAEs). Participants will also wear a Fitbit activity tracker (Inspire 3 or similar) for the duration of the study and install the Fitbit app on their smartphone. The Fitbit is a wristwatch-sized waterproof device that assesses heart and breathing rates, physical activity, and sleep, skin temperature, and oxygen levels and wirelessly transmits data to the server. Data from the wearable devices along with electronic patient-reported outcomes will be used to detect and triage immune-related adverse events.
  Interventions: Behavioral: Digital remote monitoring intervention
- Usual care (Active Comparator): This group will complete baseline, midpoint, and end of study measures and complete the Short Physical Performance Battery (SPPB) as feasible but will not wear an activity tracker or rate weekly symptoms.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Digital remote monitoring intervention — Responses to the PRO-CTCAE questions range from 0-4. Any grade 2-4 response (reflecting moderate to severe symptoms) will trigger a recommendation that the participant may want to contact their provider about the potentially concerning symptom. Fitbit data points exceeding prespecified thresholds based on physiological norms (for skin temperature and pulse oxygenation) or each participants' historic average (heart rate and activity) will also trigger a recommendation that the participant may want to contact their provider about the potentially concerning data point. Participants will receive weekly data reports that show summaries/graphs of recent alerts triggered, symptom ratings, and Fitbit data.
  Arms: Digital remote monitoring group (intervention)
Other: Usual Care — Participants will complete baseline, midpoint, and end of study measures and complete the Short Physical Performance Battery (SPPB). They will not complete surveys, wear a Fitbit, or receive recommendations about when they might want to reach out to a provider about potentially concerning symptoms or Fitbit values. Participants will use the standard information they receive from clinic about how to manage their symptoms and when to contact their care team.
  Arms: Usual care

SUMMARY:
The goal of this study is to evaluate the feasibility of using information from wearable devices and self-reported symptoms to remotely monitor patients during immunotherapy. The main questions it aims to answer are:

* Is the digital remote patient monitoring tool feasible and acceptable to patients?
* Do the alerts and guidance improve symptom management, quality of life, and engagement with the care team during treatment?

Participants will:

* Complete a demographic questionnaire at the beginning of the study and quality-of-life and health questionnaires at the beginning, midpoint, and end of study.
* As feasible: At the beginning and end of the study, complete an in-person physical function assessment measuring balance (Short Physical Performance Battery).

If participant is randomly assigned to the intervention group, they will also:

* Complete weekly symptom ratings via digital remote patient monitoring tool
* Wear a Fitbit activity tracker for 90 days.
* At the end of the study, complete a semi-structured interview to provide feedback on the study.

DETAILED DESCRIPTION:
Participants (n = 40) will be recruited from UPMC Hillman clinics.

If eligible patients consent to participate, they will complete online baseline, midpoint, and end of study questionnaires. Participant's medical records will be reviewed to extract demographic information and clinical covariates, including information about their cancer, its treatment, biological variables such as sex and age, clinical variables such as comorbidities, surgeries and hospitalizations, medications, and other markers of health care utilization (e.g., emergency department visits). Once extracted, these values will be linked only to their study ID number.

As feasible, participants will complete the Short Physical Performance Battery (SPPB) at the UPMC Hillman Cancer Center or the research team's office at baseline and at the end of the study. During these visits, this in-person assessment will be administered by trained study team members. Participants that enroll in the study remotely will be invited to complete the in-person SPPB as feasible. The SPPB will be conducted within 2 weeks of the enrollment date and within 2 weeks of the end of study date.

Following informed consent and completing baseline questionnaires, participants will then be randomized into the digital remote monitoring group or usual care (1:1).

For participants in the intervention condition (digital remote monitoring group):

At the initial study visit, participants in the digital remote monitoring group will be oriented to the ecological momentary assessment procedures to assess patient reported symptoms.

Participants in the digital remote monitoring group will receive a weekly text message containing a secure link to a brief (approximately 5 minute) online symptom survey administered via Qualtrics. Each participant is assigned a unique, non-identifying study ID, which is embedded in their survey link to ensure responses are associated with the correct participant. A secure Qualtrics-based contact log, accessible only to authorized study personnel, will maintain phone numbers and study IDs for survey distribution. No survey data is stored on the participant's device, and no personally identifiable information is collected within the survey. All data is linked only to the study ID. Data usage requirements are not significantly different from what most smartphone users would require if they use their device to access the Internet for web searching.

Symptoms will be assessed using the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). The PRO-CTCAE includes 22 symptoms commonly associated with immune-related adverse events (irAEs), such as fatigue, diarrhea, abdominal pain, constipation, rash, itchy skin, dry skin, muscle aches, joint pain, arm or leg swelling, decreased appetite, nausea, vomiting, shortness of breath, cough, headache, dry mouth, blurry vision, dizziness, pain or burning with urination, eye irritation (e.g., itching, watering, stinging, foreign body sensation), and nasal congestion. Participants are asked to report on symptoms experienced over the past 7 days. Responses are rated on a 0-4 scale.

If a participant reports a rating of 2 (moderate), 3 (severe), or 4 (very severe) for any symptom, an automated alert will appear at the end of the survey. This alert will inform participants that their responses may be concerning and that they should consider contacting their clinical care team. The alert will also include a summary of the self-reported severity, frequency, and/or interference for the relevant symptom(s), along with links to symptom management resources on the National Cancer Institute website.

In addition to the PRO-CTCAE questions in the weekly survey, participants in the digital remote monitoring group will also be asked to rate their overall quality of life for that day from 0 (worst possible) to 10 (best possible), report any cancer treatment they've received since the last survey, and indicate if they have communicated with their cancer care team since their last survey.

Participants in the digital remote monitoring group will receive weekly email reports from the study team that show summaries/graphs of recent alerts triggered, symptom ratings, and Fitbit data. Participants may choose to share these data reports with their care team, family members, etc.

Participants in the remote monitoring group will also be asked to wear a Fitbit device as feasible (Fitbit Inspire 3 or similar) for the duration of the study and to install the Fitbit app on their smartphone. The Fitbit is a wristwatch-sized waterproof device that assesses heart and breathing rates, physical activity, and sleep, skin temperature, and oxygen levels and wirelessly transmits data to the server. Participants will be asked to charge the device as needed, approximately every 4-5 days. If participants already own a Fitbit device that collects comparable data to the study provided device, the study team will request access to the participant's Fitbit data for the duration of their study participation. Fitbit data points exceeding prespecified thresholds based on physiological norms (for skin temperature and pulse oxygenation) or each participants' historic average (heart rate and activity) will trigger a recommendation that the participant may want to contact their provider about the potentially concerning data point(s).

At the end of the study, participants will complete an end of study interview.

ELIGIBILITY:
Inclusion Criteria:

* within one week of starting immune checkpoint inhibitor therapy at UPMC Hillman Cancer Center for advanced melanoma;
* age 18 years or older;
* ability to read and write in English;
* owns and uses a smartphone capable of running study applications

Exclusion Criteria:

* under 18 years old; and
* unable to read and write in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability via semi-structured interviews | At the end of the intervention (at approximately 90 days)
  Post-intervention semi-structured interviews will be conducted to gather participant feedback and assess acceptability of the intervention. Participants will be asked to rate the likelihood they would keep using system on their own and to recommend system on a scale from 0 (not at all likely) to 10 (extremely likely). Responses will be averaged.
Acceptability via System Usability Scale | At the end of the intervention (at approximately 90 days)
  System Usability Scale (SUS). For odd items, subtract one from the user response. For even-numbered items, subtract the user responses from 5. This scales all values from 0 to 4 (with four being the most positive response). Add up the converted responses for each user and multiply that total by 2.5. Possible range of scores is 0 to 100 representing a composite measure of the overall usability of the system being studied.
Feasibility via accrual rate | From enrollment to the end of the intervention (at approximately 90 days)
  accrual rate (number of participants that enroll [consent and provide at least one form of data] out of number of participants approached)
Feasibility via engagement with surveys | From enrollment to the end of the intervention (at approximately 90 days)
  engagement (how many weeks participants completed symptom surveys)
Feasibility via engagement with Fitbit | From enrollment to the end of the intervention (at approximately 90 days)
  engagement (how many days within the study the participants had Fitbit data)
Feasibility via completion rate | From enrollment to the end of the intervention (at approximately 90 days)
  completion rate (number of participants that complete the study)

SECONDARY OUTCOMES:
Patient-Reported Physical Symptoms | Change from baseline to the end of the intervention (at approximately 90 days)
  Symptoms will be assessed using the PRO version of the Common Terminology for Adverse Events (PRO-CTCAE; Dueck et al., 2015). PRO-CTCAE questions will assess 22 symptoms commonly associated with immune-related adverse events (irAEs), such as fatigue, diarrhea, abdominal pain, constipation, rash, and itchy skin. For each symptom, participants will be asked about the severity, frequency, and/or the extent to which a symptom interfered with their activities. Participants will be asked to complete one rating per week and will report on symptoms over the past 7 days. Responses range from 0-4, with higher scores indicating more severe symptoms.

OTHER OUTCOMES:
Objective physical activity | Change from baseline to the end of the intervention (at approximately 90 days)
  A Bluetooth enabled activity monitor worn throughout the study will estimate number of steps/day.
Self-Efficacy for Managing Symptoms | Change from baseline to the end of the intervention (at approximately 90 days)
  PROMIS Self-Efficacy for Managing Symptoms v1.0 - Short Form 4a is a 4-item short form assessing confidence to manage/control symptoms, to manage symptoms in different settings and to keep symptoms from interfering with work, sleep, relationships, or recreational activities. Responses are rated on a 5-point Likert scale, yielding a total score range of 4 to 16. Higher scores indicate greater perceived self-efficacy for managing symptoms.
Short Physical Performance Battery (SPPB) | Change from baseline to the end of the intervention (at approximately 90 days)
  The SPPB is a short battery of performance tests of lower extremity functioning. The tests measure gait speed, standing balance, and lower extremity strength and power. To test gait speed, patients are instructed to walk an 8-foot walking course at their usual pace with assistive devices if needed. Four progressively more challenging positions are used to test balance (bipedal [feet next to each other], semi-tandem [one foot slightly in front of the other], and full tandem [one foot in front of the other]). To test lower extremity strength, patients are asked to stand up and sit down five times as quickly as possible and are timed from the initial sitting position to the final standing position at the end of the fifth stand. Each component (gait speed, balance, chair stands) is scored 0-4, where 0 is unable to complete task and 4 indicates highest level of performance. Total score is 0-12 with higher scores indicating better lower extremity function.
Patient-Centered Communication Questionnaire - Cancer | Change from baseline to the end of the intervention (at approximately 90 days)
  The PCC-Ca-36 is a 36-item questionnaire to assess patients' experience with patient-centered communication during cancer care. It evaluates 6 core functions: exchanging information, fostering healing relationships, making decisions, attention to emotions, taking care of yourself, and dealing with uncertainty. Responses are rated on a 5-point Likert scale (1-5 with higher scores representing better communication) with some items having the option "Does not apply". Each PCC core function is scored by averaging items within the function, and an overall PCC score is the average of all items. The six core function scores and the total score range from 1-5, with higher scores indicating better perceived patient-centered communication.
Functional Assessment of Cancer Therapy - Immune Checkpoint Modulator | Change from baseline to the end of the intervention (at approximately 90 days)
  The Functional Assessment of Cancer Therapy - Immune Checkpoint Modulator (FACT-ICM) a collection of short forms assessing physical well-being, emotional well-being, social/family well-being, and functional well-being, along with immune-related treatment concerns specific to immune checkpoint modulators. Responses are rated on a 5-point Likert scale yielding a total score ranging from 0-208. A higher total score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Carissa A Low, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Preliminary IPD data from this pilot study will not be shared